CLINICAL TRIAL: NCT01122849
Title: Exploratory Subjective Sleep Study of a Prototype Nasal Dilator
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B3570674
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-01

CONDITIONS: Sleep Disorders; Congestion, Nasal
Keywords: trouble with sleep; night time nasal congestion
MeSH Terms: conditions — Sleep Wake Disorders; Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prototype Nasal Dilator (Experimental): Prototype Nasal Dilator
  Interventions: Device: Prototype Nasal Dilator
- Marketed Nasal Strip (Active Comparator): Marketed Nasal Strip
  Interventions: Device: Marketed Nasal Strip
- Placebo Nasal Strip (Placebo Comparator): Placebo
  Interventions: Device: Placebo Nasal Strip

INTERVENTIONS:
Device: Prototype Nasal Dilator — Prototype nasal dilator AB2R11
  Arms: Prototype Nasal Dilator
Device: Marketed Nasal Strip — Breathe Right Nasal Strip- Clear small/medium
  Arms: Marketed Nasal Strip
Device: Placebo Nasal Strip — Placebo strip
  Arms: Placebo Nasal Strip

SUMMARY:
The purpose of this exploratory study is to evaluate the subjective measures of congestion and sleep quality in subjects who suffer from chronic nasal congestion and report trouble with their sleep.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with leptorrhine noses
* Subjects suffering from chronic nocturnal nasal congestion and report trouble with sleep

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-10-01; Primary Completion 2010-02-01 (Actual); Study Completion 2010-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - TKL Research Inc, Paramus, New Jersey
  - Valley Clinical Research Center, Bethlehem, Pennsylvania

REFERENCES:
- [Derived] Schenkel EJ, Ciesla R, Shanga GM. Effects of nasal dilator strips on subjective measures of sleep in subjects with chronic nocturnal nasal congestion: a randomized, placebo-controlled trial. Allergy Asthma Clin Immunol. 2018 Aug 27;14:34. doi: 10.1186/s13223-018-0258-5. eCollection 2018. PMID 30154874

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at two centers in USA.
Pre-assignment Details: A total of 97 participants were screened for this study, out of which 61 participants were randomized to the study and 36 participants did not meet study criteria.
Groups:
- Marketed Nasal Strip: Participants applied the Marketed nasal strips according to written instructions. A member of the site staff reviewed the instructions for administration with each participant. Strips were applied every night during the treatment phase of the study. All treatments in this study were self-administered by the participant.
- Placebo Nasal Strip: Participants applied the Placebo nasal strips according to written instructions. A member of the site staff reviewed the instructions for administration with each participant. Strips were applied every night during the treatment phase of the study. All treatments in this study were self-administered by the participant.
- Prototype Nasal Strip: Participants applied the Prototype nasal strips according to written instructions. A member of the site staff reviewed the instructions for administration with each participant. Strips were applied every night during the treatment phase of the study. All treatments in this study were self-administered by the participant.
Period: Overall Study
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Started | 20 | 21 | 20
Completed | 20 | 21 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prototype Nasal Strip: Participants applied the Prototype nasal dilator strips according to written instructions. A member of the site staff reviewed the instructions for administration with each participant. Strips were applied every night during the treatment phase of the study. All treatments in this study were self-administered by the participant.
- Total: Total of all reporting groups
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip | Total
Number analyzed (Participants) | 20 | 21 | 20 | 61
Age, Customized [Mean (Standard Deviation); unit: Years]
  Years | 46.1 (10.17) | 44.5 (9.59) | 42.5 (13.97) | 44.4 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 15 | 50
  Male | 2 | 4 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 20 | 21 | 20 | 61
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Average Score Using Pittsburgh Insomnia Rating Scale (PIRS) in Q1, Q3, Q17 and Q18 at Day 7
Description: The PIRS questionnaire had 3 sections (Section A [Q1 to Q12], Section B [Q13 to 16] and Section C [Q17 to Q20]). The following questions were asked from Section A : 1. One or more awakenings after getting to sleep and 3 Sleep that does not fully refresh you, and Section C: 17 Your sleep quality compared to most people and 18 Your satisfaction with your sleep. Section A question were scored as follows: 0= Not at all bothered, 1= slightly bothered, 2=moderately bothered, and 3= severely bothered. Section B, Q13 and 14 were scored as follows 0= Less than ½ hour, 1= between ½ to 1 hour, 2= between 1 to 3 hours and 3=more than 3 hours or I didn't sleep; Q15 and 16 were scored as 0=more than 7 hours, 1= between 4 to 7 hours, 2= between 2 to 4 hours, and 3=Less than 2 hours or I didn't sleep. Section C questions were scored as follows: 0=Excellent, 1=Good, 2=Fair, and 3=Poor. Lower PIRS score shows better sleep quality.
Time Frame: At Baseline and Day 7
Population: Analysis for this outcome was performed on intent-to-treat (ITT) population, defined as all participants who were randomized and had at least one post-baseline efficacy assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a scale
  Q1 | -0.911 [-1.21 to -0.61] | -0.694 [-0.99 to -0.40] | -1.032 [-1.34 to -0.72]
  Q3 | -1.004 [-1.37 to -0.63] | -0.708 [-1.07 to -0.34] | -0.947 [-1.33 to -0.56]
  Q17 | -0.721 [-1.01 to -0.43] | -0.349 [-0.63 to -0.07] | -0.539 [-0.84 to -0.24]
  Q18 | -0.643 [-0.91 to -0.38] | -0.234 [-0.50 to 0.03] | -0.697 [-0.98 to -0.42]
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison of Q1 at Day 7; Test type: Superiority or Other; p = 0.5456, ANCOVA — Between treatment p-values and confidence intervals; Least Square (LS) Mean difference = -0.12, 95% CI 2-sided [-0.52 to 0.28]
Statistical Analysis 2: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison of Q1 at Day 7; Test type: Superiority or Other; p = 0.1029, ANCOVA — Between treatment p-values and confidence intervals; LS mean difference = -0.34, 95% CI 2-sided [-0.75 to 0.07]
Statistical Analysis 3: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison of Q1 at Day 7; Test type: Superiority or Other; p = 0.2879, ANCOVA — Between treatment p-values and confidence intervals; LS mean difference = 0.22, 95% CI 2-sided [-0.19 to 0.62]
Statistical Analysis 4: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison for Q3 at Day 7; Test type: Superiority or Other; p = 0.8213, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 0.06, 95% CI 2-sided [-0.45 to 0.56]
Statistical Analysis 5: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison for Q3 at Day 7; Test type: Superiority or Other; p = 0.3457, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = -0.24, 95% CI [-0.74 to 0.27]
Statistical Analysis 6: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison for Q3 at Day 7; Test type: Superiority or Other; p = 0.2364, ANCOVA; LS Mean Difference = 0.30, 95% CI 2-sided [-0.20 to 0.79]
Statistical Analysis 7: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison for Q17 at Day 7; Test type: Superiority or Other; p = 0.3553, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 0.18, 95% CI 2-sided [-0.21 to 0.57]
Statistical Analysis 8: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison for Q17 at Day 7; Test type: Superiority or Other; p = 0.3369, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -0.19, 95% CI 2-sided [-0.58 to 0.20]
Statistical Analysis 9: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison for Q17 at Day 7; Test type: Superiority or Other; p = 0.0591, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 0.37, 95% CI 2-sided [-0.01 to 0.76]
Statistical Analysis 10: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison of Q18 at Day 7; Test type: Superiority or Other; p = 0.7686, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -0.05, 95% CI 2-sided [-0.42 to 0.31]
Statistical Analysis 11: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison of Q18 at Day 7; Test type: Superiority or Other; p = 0.0151, ANCOVA; LS Mean Difference = -0.46, 95% CI 2-sided [-0.83 to -0.09]
Statistical Analysis 12: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison of Q18 at Day 7; Test type: Superiority or Other; p = 0.0256, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 0.41, 95% CI 2-sided [0.05 to 0.77]

2. Primary Outcome: Change From Baseline in Mean Average Score Using Pittsburgh Insomnia Rating Scale (PIRS) in Q1, Q3, Q17 and Q18 at Day 14
Description: Participant were asked questions related to their sleep using PIRS questionnaire. The PIRS questionnaire had 3 sections. Section A (Q1 to Q12), Section B (Q13 to Q16) and Section C (Q17 to Q20). Section A question were scored as follows: 0= Not at all bothered, 1= slightly bothered, 2=moderately bothered, and 3= severely bothered. Section B questions 13 and 14 were scored as follows 0= Less than ½ hour, 1= between ½ to 1 hour, 2= between 1 to 3 hours and 3=more than 3 hours or I didn't sleep; Questions 15 and 16 were scored as 0=more than 7 hours, 1= between 4 to 7 hours, 2= between 2 to 4 hours, and 3=Less than 2 hours or I didn't sleep. Section C questions were scored as follows: 0=Excellent, 1=Good, 2=Fair, and 3=Poor. Lower PIRS score shows better sleep quality.
Time Frame: At Baseline and Day 14
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- Marketed Nasal Strip: Participants applied the Marketed nasal strips according to written instructions. A member of the site staff reviewed the instructions for administration with each participant. The strips were applied every night during the treatment phase of the study. All treatments in this study were self-administered by the participant.
- Placebo Nasal Strip: Participants applied the Placebo nasal strips according to written instructions. A member of the site staff reviewed the instructions for administration with each participant. The strips were applied every night during the treatment phase of the study. All treatments in this study were self-administered by the participant.
- Prototype Nasal Strip: Participants applied the Prototype nasal strips according to written instructions. A member of the site staff reviewed the instructions for administration with each participant. The strips were applied every night during the treatment phase of the study. All treatments in this study were self-administered by the participant.
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a scale
  Q1 (One or more awakenings after getting to sleep) | -1.047 [-1.36 to -0.74] | -0.844 [-1.14 to -0.54] | -1.157 [-1.48 to -0.84]
  Q3 (Sleep that does not fully refresh you) | -1.306 [-1.69 to -0.92] | -0.917 [-1.30 to -0.54] | -1.104 [-1.50 to -0.70]
  Q17 (Your sleep quality compared to most people) | -0.714 [-1.04 to -0.39] | -0.359 [-0.68 to -0.04] | -0.837 [-1.17 to -0.50]
  Q18 (Your satisfaction with your sleep) | -0.873 [-1.18 to -0.57] | -0.464 [-0.76 to -0.16] | -0.951 [-1.27 to -0.63]
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison of Q1at Day 14; Test type: Superiority or Other; p = 0.5958, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -0.11, 95% CI 2-sided [-0.52 to 0.30]
Statistical Analysis 2: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison of Q1 at Day 14; Test type: Superiority or Other; p = 0.1429, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -0.31, 95% CI 2-sided [-0.73 to 0.11]
Statistical Analysis 3: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison of Q1 at Day 14; Test type: Superiority or Other; p = 0.3348, ANCOVA; LS Mean Difference = 0.20, 95% CI 2-sided [-0.21 to 0.62]
Statistical Analysis 4: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison of Q3 at Day 14; Test type: Superiority or Other; p = 0.4425, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 0.20, 95% CI [-0.32 to 0.72]
Statistical Analysis 5: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison of Q3 at Day 14; Test type: Superiority or Other; p = 0.4795, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.71 to 0.34]
Statistical Analysis 6: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison of Q3 at Day 14; Test type: Superiority or Other; p = 0.1375, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 0.39, 95% CI 2-sided [-0.13 to 0.90]
Statistical Analysis 7: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison of Q17 at Day 14; Test type: Superiority or Other; p = 0.5750, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -0.12, 95% CI 2-sided [-0.56 to 0.31]
Statistical Analysis 8: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison of Q17 at Day 14; Test type: Superiority or Other; p = 0.0337, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -0.48, 95% CI 2-sided [-0.92 to -0.04]
Statistical Analysis 9: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison of Q17 at Day 14; Test type: Superiority or Other; p = 0.1061, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 0.35, 95% CI 2-sided [-0.08 to 0.79]
Statistical Analysis 10: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison of Q18 at Day 14; Test type: Superiority or Other; p = 0.7092, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -0.08, 95% CI 2-sided [-0.50 to 0.34]
Statistical Analysis 11: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison of Q18 at Day14; Test type: Superiority or Other; p = 0.0250, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = -0.49, 95% CI 2-sided [-0.91 to -0.06]
Statistical Analysis 12: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison for Q18 at Day 14; Test type: Superiority or Other; p = 0.0503, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 0.41, 95% CI 2-sided [0.00 to 0.82]

3. Primary Outcome: Change From Baseline in Mean Average Score of NRQLQ (Nocturnal Rhino Conjunctivitis Quality of Life Questionnaire) for Each Domain (Sleep, Sleep Time, Symptoms on Waking in the Morning, and Practical Problems) on the) at Day 7
Description: Participants scored all the domains of NRQLQ using same 7 points scale where 0=Not troubled and 6=extremely troubled. Sleep problems (difficulty getting sleep, unable to get a good night sleep or wake up during the night, restless [tossing and turning] and having to get up because stuffy nose or to blow nose using the score, scores range: Min-Max [0-24]), Sleep time problems (Nasal congestion or stuffy nose, sinus pressure or pain, runny nose, post-nasal drip [drainage down back of nose/throat], and headache, scores range: 0-30); Symptoms on waking in the morning (Feel tired and unrefreshed, nasal congestion or stuffy nose, congestion in sinuses, takes time to clear nighttime drainage after waking up, scores range:0-24); practical problems (have to avoid symptom triggers (such as dust, cigarette smoke, strong smells and perfumes, need to rub nose or eyes, and have to take medication, scores range: 0-18). Lower scores indicate improvement in the rhinitis symptoms.
Time Frame: At Baseline and Day 7
Population: Analysis for this outcome was performed on ITT population, defined as all participants who were randomized and had at least one post-baseline efficacy assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a Scale
  Sleep Problems | -7.398 [-9.44 to -5.36] | -4.194 [-6.18 to -2.21] | -6.563 [-8.71 to -4.42]
  Sleep time Problems | -7.494 [-9.99 to -5.00] | -5.638 [-8.09 to -3.19] | -8.212 [-10.81 to -5.61]
  Symptoms on walking in the morning | -7.196 [-9.28 to -5.11] | -4.074 [-6.13 to -2.02] | -7.905 [-10.09 to -5.72]
  Practical Problems | -2.774 [-4.02 to -1.52] | -2.277 [-3.51 to -1.04] | -3.079 [-4.38 to -1.78]
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison for sleep problems at Day 7; Test type: Superiority or Other; p = 0.5462, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 0.84, 95% CI 2-sided [-1.92 to 3.59]
Statistical Analysis 2: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison for sleep problems at Day 7; Test type: Superiority or Other; p = 0.0942, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -2.37, 95% CI 2-sided [-5.16 to 0.42]
Statistical Analysis 3: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison of sleep problems at Day 7; Test type: Superiority or Other; p = 0.0221, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 3.20, 95% CI 2-sided [0.48 to 5.93]
Statistical Analysis 4: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison of Sleep Time problems at Day 7; Test type: Superiority or Other; p = 0.6731, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = -0.72, 95% CI 2-sided [-4.11 to 2.68]
Statistical Analysis 5: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison for Sleep time problems at Day 7; Test type: Superiority or Other; p = 0.1354, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -2.57, 95% CI 2-sided [-5.98 to 0.83]
Statistical Analysis 6: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison of sleep time problems at Day 7; Test type: Superiority or Other; p = 0.2722, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = 1.86, 95% CI 2-sided [-1.50 to 5.21]
Statistical Analysis 7: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison for symptoms on walking in the morning at Day 7; Test type: Superiority or Other; p = 0.6195, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = -0.71, 95% CI 2-sided [-3.55 to 2.14]
Statistical Analysis 8: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison at day 7 for symptoms for walking in the morning; Test type: Superiority or Other; p = 0.0099, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -3.83, 95% CI 2-sided [-6.70 to -0.96]
Statistical Analysis 9: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison for symptoms on waking in the morning at Day 7; Test type: Superiority or Other; p = 0.0298, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 3.12, 95% CI 2-sided [0.32 to 5.93]
Statistical Analysis 10: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison for practical problems at Day 7; Test type: Superiority or Other; p = 0.7211, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = -0.30, 95% CI 2-sided [-2.01 to 1.40]
Statistical Analysis 11: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison for practical problems at Day 7; Test type: Superiority or Other; p = 0.3500, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = -0.80, 95% CI 2-sided [-2.51 to 0.90]
Statistical Analysis 12: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison for practical problems at Day 7; Test type: Superiority or Other; p = 0.5564, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = 0.50, 95% CI 2-sided [-1.19 to 2.18]

4. Primary Outcome: Change From Baseline in Mean Average Score of NRQLQ (Nocturnal Rhino Conjunctivitis Quality of Life Questionnaire) for Each Domain (Sleep, Sleep Time, Symptoms on Waking in the Morning, and Practical Problems) on the) at Day 14
Description: Participants scored all the domains of NRQLQ using same 7 points scale where 0=Not troubled and 6=extremely troubled. Sleep problems (difficulty getting sleep, unable to get a good night sleep or wake up during the night, restless [tossing and turning] and having to get up because stuffy nose or to blow nose using the score, scores range: Min-Max [0-24]), Sleep time problems (Nasal congestion or stuffy nose, sinus pressure or pain, runny nose, post-nasal drip [drainage down back of nose/throat], and headache, scores range: 0-30); Symptoms on waking in the morning (Feel tired and unrefreshed, nasal congestion or stuffy nose, congestion in sinuses, takes time to clear nighttime drainage after waking up, scores range:0-24); practical problems (have to avoid symptom triggers such as dust, cigarette smoke, strong smells and perfumes, need to rub nose or eyes, and have to take medication, scores range: 0-18). Lower scores indicate improvement in the rhinitis symptoms.
Time Frame: At Baseline and Day 14
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a scale
  Sleep Problems | -7.624 [-9.68 to -5.57] | -5.738 [-7.74 to -3.74] | -7.051 [-9.21 to -4.89]
  Sleep Time Problems | -8.746 [-11.24 to -6.26] | -7.051 [-9.49 to -4.61] | -6.768 [-9.36 to -4.18]
  Symptoms on waking in the morning | -7.858 [-9.90 to -5.81] | -5.318 [-7.33 to -3.30] | -8.001 [-10.14 to -5.86]
  Practical Problems | -3.591 [-4.74 to -2.44] | -3.208 [-4.34 to -2.07] | -3.054 [-4.25 to -1.86]
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison for Sleep Problems at Day 14; Test type: Superiority or Other; p = 0.6804, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 0.57, 95% CI 2-sided [-2.20 to 3.35]
Statistical Analysis 2: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison for sleep problems at Day 14; Test type: Superiority or Other; p = 0.3524, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -1.31, 95% CI 2-sided [-4.12 to 1.49]
Statistical Analysis 3: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison for sleep problems at Day 14; Test type: Superiority or Other; p = 0.1739, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 1.89, 95% CI 2-sided [-0.86 to 4.63]
Statistical Analysis 4: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison for Sleep time problems at Day 14; Test type: Superiority or Other; p = 0.2463, ANCOVA — Between treatment p-values and confidence intervals; Between treatment p-values and confidence intervals; LS Mean difference = 1.98, 95% CI 2-sided [-1.41 to 5.36]
Statistical Analysis 5: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison for sleep time problems at Day 14; Test type: Superiority or Other; p = 0.8677, ANCOVA; LS Mean difference = 0.28, 95% CI 2-sided [-3.11 to 3.68]
Statistical Analysis 6: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison for sleep time problems at Day 14; Test type: Superiority or Other; p = 0.3136, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 1.70, 95% CI 2-sided [-1.65 to 5.04]
Statistical Analysis 7: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison for symptoms on waking in the morning at Day 14; Test type: Superiority or Other; p = 0.9183, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -0.14, 95% CI 2-sided [-2.93 to 2.65]
Statistical Analysis 8: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison for symptoms on waking in the morning at Day 14; Test type: Superiority or Other; p = 0.0614, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = -2.68, 95% CI 2-sided [-5.50 to 0.13]
Statistical Analysis 9: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison for symptoms on waking in the morning at Day 14; Test type: Superiority or Other; p = 0.0695, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 2.54, 95% CI 2-sided [-0.21 to 5.29]
Statistical Analysis 10: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison for practical problems at Day14; Test type: Superiority or Other; p = 0.4947, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = 0.54, 95% CI 2-sided [-1.03 to 2.10]
Statistical Analysis 11: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison for practical problems at Day 14; Test type: Superiority or Other; p = 0.8454, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = 0.15, 95% CI 2-sided [-1.42 to 1.72]
Statistical Analysis 12: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison for practical problems at Day 14; Test type: Superiority or Other; p = 0.6223, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = 0.38, 95% CI 2-sided [-1.17 to 1.93]

5. Primary Outcome: Change From Baseline in Mean Sum of 7 Questions of Congestion Quantifier 7 Questionnaire (CQ7) at Day 7
Description: Participants answered following questions of CQ7 questionnaire: Q1 -How often did you have nasal stuffiness, blockage, or congestion?, Q2- How often did you have sinus pressure or pain in your face?, Q3-How often did you have to breathe through your mouth because you could not breathe through your nose?, Q4-How often did you have difficulty completely clearing your nose even after repeated blowing?, Q5-How often did any of these symptoms affect your ability to work, learn in school, or do the things you need to do?, Q6-How often did you awaken in the morning with nasal stuffiness, blockage, or congestion?, Q7-How often was your sleep affected by your nasal stuffiness, blockage, or congestion?. Their responses were scored using a 5 point scale where 0=none of the time; 1=a little of the time, 2=some of the time, 3=most of the time, 4=all of the time. Lower CQ7 scores reflect better nasal patency.
Time Frame: At Baseline and Day 7
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a scale | -6.845 [-9.28 to -4.41] | -5.137 [-7.53 to -2.74] | -8.184 [-10.75 to -5.62]
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison at Day 7; Test type: Superiority or Other; p = 0.4258, LS Mean Difference — Between treatment p-values and confidence intervals; LS Mean difference = -1.34, 95% CI 2-sided [-4.68 to 2.01]
Statistical Analysis 2: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison at Day 7; Test type: Superiority or Other; p = 0.0764, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -3.05, 95% CI 2-sided [-6.43 to 0.33]
Statistical Analysis 3: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison at Day 7; Test type: Superiority or Other; p = 0.2986, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 1.71, 95% CI 2-sided [-1.56 to 4.97]

6. Primary Outcome: Change From Baseline in Mean Sum of 7 Questions of Congestion Quantifier 7 Questionnaire (CQ7) at Day 14
Description: Participants answered following questions of CQ7 questionnaire: Q1 -How often did you have nasal stuffiness, blockage, or congestion?, Q2- How often did you have sinus pressure or pain in your face?, Q3-How often did you have to breathe through your mouth because you could not breathe through your nose?, Q4-How often did you have difficulty completely clearing your nose even after repeated blowing?, Q5-How often did any of these symptoms affect your ability to work, learn in school, or do the things you need to do?, Q6-How often did you awaken in the morning with nasal stuffiness, blockage, or congestion?, Q7-How often was your sleep affected by your nasal stuffiness, blockage, or congestion?. Their responses were scored using a 5 point scale where 0=none of the time; 1=a little of the time, 2=some of the time, 3=most of the time, 4=all of the time. Lowe CQ7 scores reflect better nasal patency.
Time Frame: At Baseline and Day 14
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a Scale | -8.035 [-10.34 to -5.73] | -5.102 [-7.37 to -2.83] | -6.917 [-9.35 to -4.49]
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Test type: Superiority or Other; p = 0.4820, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 1.12, 95% CI 2-sided [-2.05 to 4.29]
Statistical Analysis 2: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Test type: Superiority or Other; p = 0.2607, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -1.81, 95% CI 2-sided [-5.02 to 1.39]
Statistical Analysis 3: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Test type: Superiority or Other; p = 0.0623, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 2.93, 95% CI 2-sided [-0.16 to 6.02]

7. Primary Outcome: Mean Score in Response to Daily Diary VAS Scale Questions Before and After Strip Application at Bedtime on Day 7
Description: Participants were asked how easy it was to breathe through their nose before and after strip application at bedtime. The participants scored their responses on 100 point VAS scale where 0 = extremely difficult to breathe and 100 = extremely easy to breathe. These responses were recorded daily.
Time Frame: Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 19 | 19
Score on scale
  Before strip application | 32.10 (22.386) | 36.37 (21.945) | 40.53 (18.234)
  After strip application | 58.95 (28.543) | 47.42 (26.742) | 61.11 (21.787)
  Change from Baseline | 23.25 (72.4) | 8.75 (24.0) | 18.89 (46.6)
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Test type: Superiority or Other; p = 0.5278, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -4.36, 95% CI 2-sided [-18.1 to 9.39]
Statistical Analysis 2: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Test type: Superiority or Other; p = 0.1458, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 10.14, 95% CI 2-sided [-3.64 to 23.93]
Statistical Analysis 3: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Test type: Superiority or Other; p = 0.0370, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -14.50, 95% CI 2-sided [-28.1 to -0.91]

8. Primary Outcome: Mean Score in Response to Daily Diary VAS Scale Questions Before and After Strip Application at Bedtime on Day 14
Description: as for outcome 7
Time Frame: Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a scale
  Before strip application: number analyzed (Participants) | 20 | 19 | 18
  Before strip application | 39.90 (24.070) | 43.21 (24.001) | 45.89 (22.292)
  After strip application: number analyzed (Participants) | 20 | 20 | 18
  After strip application | 68.70 (26.636) | 51.05 (25.387) | 67.56 (23.605)
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Test type: Superiority or Other; p = 0.4483, ANCOVA; Between treatment p-values and confidence intervals; LS Mean Difference = -5.10, 95% CI 2-sided [-18.5 to 8.29]
Statistical Analysis 2: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Test type: Superiority or Other; p = 0.0385, ANCOVA; Between treatment p-values and confidence intervals; LS Mean Difference = 14.28, 95% CI 2-sided [0.79 to 27.77]
Statistical Analysis 3: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Test type: Superiority or Other; p = 0.0046, ANCOVA; Between treatment p-values and confidence intervals; LS Mean difference = -19.37, 95% CI 2-sided [-32.5 to -6.23]

9. Primary Outcome: Mean Score in Response to Daily Diary VAS Scale Questions Before and After Strip Removal in Morning on Day 7
Description: Participants were asked how easy it was to breathe through their nose before and after strip removal in morning. The participants scored their responses on 100 point VAS scale where 0 = extremely difficult to breathe and 100 = extremely easy to breathe. These responses were recorded daily.
Time Frame: Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a Scale
  Before strip removal | 60.15 (25.522) | 46.95 (25.888) | 62.63 (19.774)
  After strip removal: number analyzed (Participants) | 20 | 19 | 19
  After strip removal | 43.10 (21.711) | 44.74 (25.236) | 60.00 (21.654)
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Test type: Superiority or Other; p = 0.0029, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 15.24, 95% CI 2-sided [5.45 to 25.02]
Statistical Analysis 2: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Test type: Superiority or Other; p = 0.4683, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 3.74, 95% CI 2-sided [-6.53 to 14.01]
Statistical Analysis 3: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Test type: Superiority or Other; p = 0.0259, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 11.50, 95% CI 2-sided [1.44 to 21.55]

10. Primary Outcome: Mean Score in Response to Daily Diary VAS Scale Questions Before and After Strip Removal in Morning on Day 14.
Description: Participants were asked how easy it was to breathe through their nose before and after strip removal in morning. The participants scored their responses on 100 point VAS scale where 0=extremely difficult to breathe and 100=extremely easy
Time Frame: Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a scale
  Before Strip Removal: number analyzed (Participants) | 20 | 19 | 18
  Before Strip Removal | 67.80 (24.816) | 48.95 (26.511) | 70.61 (22.078)
  After Strip Removal: number analyzed (Participants) | 20 | 19 | 18
  After Strip Removal | 51.35 (25.203) | 45.26 (25.473) | 61.11 (21.978)
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Test type: Superiority or Other; p = 0.1764, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 7.79, 95% CI 2-sided [-3.62 to 19.19]
Statistical Analysis 2: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Test type: Superiority or Other; p = 0.9183, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 0.63, 95% CI 2-sided [-11.7 to 12.94]
Statistical Analysis 3: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Test type: Superiority or Other; p = 0.2313, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 7.16, 95% CI [-4.70 to 19.01]

11. Primary Outcome: Mean Score in Response to Daily Diary Questions (Q2 and Q4) at Bedtime on Day 7
Description: Questions regarding nasal strips were asked to participants and scores were noted on daily basis. Participants were asked how stuffed their nose felt before and after strip application (Q2) and how breathing felt after strip was applied (Q4) at bedtime. For Q2 the participants scored their responses on a scale of 0 to 3 where 0=no symptoms, 1=mild symptoms, 2=moderate symptoms, 3=severe symptoms. For Q4, participants scored their responses on a scale of -5 to 5 where -5=much worse, 0=same, and 5=much better (Q4 was asked after strip application only therefore no data for before application is available for Q4.)
Time Frame: Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Marketed Nasal Strip: Participants applied the Marketed nasal strips according to written instructions to be provided. A member of the site staff reviewed the instructions for administration with each participant. Strips were applied every night during the treatment phase of the study. All treatments in this study were self-administered by the participant.
- Placebo Nasal Strip: Participants applied the Placebo nasal strips according to written instructions to be provided. A member of the site staff reviewed the instructions for administration with each participant. Strips were applied every night during the treatment phase of the study. All treatments in this study were self-administered by the participant.
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a Scale
  Before strip application (Q2) | 1.75 (0.550) | 1.70 (0.733) | 1.63 (0.597)
  After strip application (Q2) | 1.00 (0.795) | 1.55 (0.887) | 1.16 (0.688)
  After strip application (Q4) | 2.80 (1.399) | 1.20 (1.473) | 1.79 (1.475)
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison for Q2 at Day 7; Test type: Superiority or Other; p = 0.1345, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = 0.27, 95% CI 2-sided [-0.09 to 0.63]
Statistical Analysis 2: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison for Q2 at Day 7; Test type: Superiority or Other; p = 0.0815, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -0.32, 95% CI 2-sided [-0.68 to 0.04]
Statistical Analysis 3: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison for Q2 at Day 7; Test type: Superiority or Other; p = 0.0015, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 0.59, 95% CI 2-sided [0.24 to 0.94]
Statistical Analysis 4: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison for Q4 at Day 7; Test type: Superiority or Other; p = 0.0292, ANCOVA — Between treatment p-values and confidence intervals; LS mean differnence = -1.03, 95% CI [-1.96 to -0.11]
Statistical Analysis 5: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison of Q4 at Day 7; Test type: Superiority or Other; p = 0.2497, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = 0.54, 95% CI 2-sided [-0.39 to 1.47]
Statistical Analysis 6: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison for Q4 at Day 7; Test type: Superiority or Other; p = 0.0011, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = -1.57, 95% CI 2-sided [-2.48 to -0.66]

12. Primary Outcome: Mean Score in Response to Daily Diary Questions (Q2 and Q4) at Bedtime on Day 14
Description: Questions regarding nasal strips were asked to participants and scores were noted on daily basis. Participants were asked how stuffed their nose felt before and after strip application (Q2) and how breathing felt after strip was applied (Q4) at bedtime. For Q2, the participants scored their responses on a scale of 0 to 3 where 0=no symptoms, 1=mild symptoms, 2=moderate symptoms, 3=severe symptoms. For Q4, participants scored their responses on a scale of -5 to 5 where -5=much worse, 0=same, and 5=much better (Q4 was asked after strip application only therefore no data for before application is available for question 4.)
Time Frame: Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a scale
  Before strip application (Q2): number analyzed (Participants) | 20 | 20 | 18
  Before strip application (Q2) | 1.40 (0.598) | 1.58 (0.607) | 1.61 (0.698)
  After strip application (Q2): number analyzed (Participants) | 20 | 17 | 18
  After strip application (Q2) | 0.85 (0.875) | 1.35 (0.786) | 1.06 (0.873)
  After strip application (Q4): number analyzed (Participants) | 20 | 20 | 18
  After strip application (Q4) | 2.70 (1.658) | 0.89 (1.410) | 2.00 (1.715)
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison for Q2 at Day 14; Test type: Superiority or Other; p = 0.8063, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 0.06, 95% CI 2-sided [-0.40 to 0.51]
Statistical Analysis 2: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison for Q2 at Day 14; Test type: Superiority or Other; p = 0.1356, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Differnence = -0.35, 95% CI 2-sided [-0.82 to 0.11]
Statistical Analysis 3: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison for Q2 at Day 14; Test type: Superiority or Other; p = 0.0786, ANCOVA; LS mean Difference = 0.41, 95% CI 2-sided [-0.05 to 0.87]
Statistical Analysis 4: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparisons for Q4 at Day 14; Test type: Superiority or Other; p = 0.1693, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -0.72, 95% CI 2-sided [-1.75 to 0.32]
Statistical Analysis 5: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison for Q4 at Day 14; Test type: Superiority or Other; p = 0.0438, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = 1.08, 95% CI 2-sided [0.03 to 2.13]
Statistical Analysis 6: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison for Q4 at Day 14; Test type: Superiority or Other; p = 0.0009, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = -1.80, 95% CI 2-sided [-2.82 to -0.78]

13. Primary Outcome: Mean Score in Response to Daily Diary Questions (Q2 and Q4) in Morning on Day 7
Description: Questions regarding nasal strips were asked to participants and scores were noted on daily basis. Participants were asked how stuffed their nose felt before and after strip removal (Q2) and how breathing felt after strip was removed (Q4) in morning. For Q2 the participants scored their responses on a scale of 0 to 3 where 0=no symptoms, 1=mild symptoms, 2=moderate symptoms, 3=severe symptoms. For Q4, participants scored their responses on a scale of -5 to 5 where -5=much worse, 0=same, and 5=much better. (Q4 was asked after strip removal only therefore no data for before removal is available for question 4.)
Time Frame: Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Prototype Nasal Strip: Participants applied the Prototype nasal strips according to written instructions to be provided. A member of the site staff reviewed the instructions for administration with each participant. Strips were applied every night during the treatment phase of the study. All treatments in this study were self-administered by the participant.
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a scale
  Before strip removal (Q2) | 1.00 (0.649) | 1.60 (0.995) | 1.00 (0.745)
  After strip removal (Q2) | 1.35 (0.671) | 1.75 (0.967) | 1.11 (0.809)
  After strip removal (Q4) | -0.20 (2.118) | 0.60 (1.759) | 1.16 (2.007)
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison for Q2 at Day 7; Test type: Superiority or Other; p = 0.1991, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = -0.24, 95% CI 2-sided [-0.62 to 0.13]
Statistical Analysis 2: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison of Q2 at Day 7; Test type: Superiority or Other; p = 0.2964, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = -0.21, 95% CI 2-sided [-0.60 to 0.19]
Statistical Analysis 3: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison of Q2 at Day 7; Test type: Superiority or Other; p = 0.8495, ANCOVA — Between treatment p-values and confidence intervals; LS mean difference = -0.04, 95% CI 2-sided [-0.42 to 0.35]
Statistical Analysis 4: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison for Q4 at Day 7; Test type: Superiority or Other; p = 0.0381, ANCOVA — Between treatment p-values and confidence intervals; LS mean difference = 1.35, 95% CI 2-sided [0.08 to 2.62]
Statistical Analysis 5: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison of Q4 at Day 7; Test type: Superiority or Other; p = 0.4005, ANCOVA — Between treatment p-values and confidence intervals; LS mean difference = 0.54, 95% CI 2-sided [-0.74 to 1.82]
Statistical Analysis 6: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison of Q4 at Day 7; Test type: Superiority or Other; p = 0.2020, ANCOVA — Between treatment p-values and confidence intervals; LS mean difference = 0.81, 95% CI 2-sided [-0.45 to 2.07]

14. Primary Outcome: Mean Score in Response to Daily Diary Questions (Q2 and Q4) in Morning on Day 14
Description: Questions regarding nasal strips were asked to participants and scores were noted on daily basis. Participants were asked how stuffed their nose felt before and after strip removal (Q2) and how breathing felt after strip was removed (Q4) in morning. For Q2 the participants scored their responses on a scale of 0 to 3 where 0=no symptoms, 1=mild symptoms, 2=moderate symptoms, 3=severe symptoms. For Q4, participants scored their responses on a scale of -5 to 5 where -5=much worse, 0=same, and 5=much better (Q4 was asked after strip removal only therefore no data for before removal is available for question 4.)
Time Frame: Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score ona scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score ona scale
  Before strip removal (Q2): number analyzed (Participants) | 20 | 20 | 18
  Before strip removal (Q2) | 0.95 (0.826) | 1.40 (0.940) | 0.89 (0.832)
  After strip removal (Q2): number analyzed (Participants) | 20 | 20 | 18
  After strip removal (Q2) | 1.30 (0.657) | 1.45 (0.887) | 1.17 (0.707)
  After strip removal (Q4): number analyzed (Participants) | 20 | 20 | 18
  After strip removal (Q4) | -0.45 (2.282) | 0.60 (1.536) | 0.94 (2.261)
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison for Q2 at Day 14; Test type: Superiority or Other; p = 0.5741, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = -0.09, 95% CI 2-sided [-0.41 to 0.23]
Statistical Analysis 2: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison for Q2 at Day 14; Test type: Superiority or Other; p = 0.6935, ANCOVA — Between treatment p-values and confidence intervals; LS Mean Difference = 0.06, 95% CI 2-sided [-0.26 to 0.39]
Statistical Analysis 3: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison of Q2 at Day 14; Test type: Superiority or Other; p = 0.3330, ANCOVA — Between treatment p-values and confidence intervals; LS mean difference = -0.15, 95% CI 2-sided [-0.47 to 0.16]
Statistical Analysis 4: Comparison: Marketed Nasal Strip vs Prototype Nasal Strip; Comparison for Q4 at Day 14; Test type: Superiority or Other; p = 0.0434, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = 1.39, 95% CI 2-sided [0.04 to 2.73]
Statistical Analysis 5: Comparison: Placebo Nasal Strip vs Prototype Nasal Strip; Comparison for Q4 at Day 14; Test type: Superiority or Other; p = 0.6333, ANCOVA — Between treatment p-values and confidence intervals; LS Mean difference = 0.32, 95% CI 2-sided [-1.02 to 1.67]
Statistical Analysis 6: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Comparison for Q4 at Day 14; Test type: Superiority or Other; p = 0.1091, ANCOVA — Between treatment p-values and confidence intervals; LS mean difference = 1.06, 95% CI 2-sided [-0.25 to 2.37]

15. Secondary Outcome: Summary for Other Questions of PIRS Questionnaire
Description: The following questions were asked from Section A (Q1 to Q12; 2 Not getting enough sleep, 4 Poor alertness during the daytime, 5 Difficulty keeping your thoughts focused, 6 Others noticing you appeared tired or fatigued, 7 too many difficulties to overcome, 8 Bad moods because you had poor sleep, 9 Lack of energy because of poor sleep, 10 Poor sleep that interferes with your relationships, 11 Being unable to sleep, 12 Being able to do only enough to get by, Section B (Q13 to Q16; 13 From the time you tried to go to sleep, How long did it take to fall asleep on most nights, 14 If you woke during the night, how long did it take to fall back to sleep on most nights,15 Not counting times when you were awake in bed, how many hours of actual sleep did you get during the worst night, 16 On how many days did you have trouble coping because of poor sleep and Section C (Q17 to Q20;, 19 The regularity of your sleep, 20 The soundness of your sleep)
Time Frame: At Day 7 and Day 14
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a Scale
  Q2 (Day 7) | 1.20 (0.894) | 1.40 (0.883) | 1.37 (0.831)
  Q2 (Day 14) | 0.90 (0.788) | 1.20 (0.834) | 0.95 (0.705)
  Q4 (Day7) | 0.75 (0.786) | 1.05 (0.945) | 0.84 (0.834)
  Q4 (Day 14) | 0.65 (0.745) | 0.90 (0.788) | 0.63 (0.684)
  Q5 (Day 7) | 0.65 (0.671) | 0.85 (0.813) | 0.63 (0.684)
  Q5 (Day 14) | 0.55 (0.605) | 0.65 (0.813) | 0.63 (0.597)
  Q6 (Day 7) | 0.50 (0.827) | 0.70 (0.923) | 0.68 (0.820)
  Q6 (Day 14) | 0.50 (0.761) | 0.60 (0.754) | 0.58 (0.692)
  Q7 (Day 7) | 0.45 (0.686) | 0.60 (0.883) | 0.37 (0.597)
  Q7 (Day 14) | 0.45 (0.826) | 0.40 (0.681) | 0.32 (0.478)
  Q8 (Day 7) | 0.65 (0.813) | 0.80 (0.894) | 0.63 (0.684)
  Q8 (Day 14) | 0.65 (0.745) | 0.55 (0.686) | 0.37 (0.597)
  Q9 (Day 7) | 0.95 (0.826) | 1.40 (0.995) | 0.89 (0.658)
  Q9 (Day 14) | 0.80 (0.834) | 0.85 (0.813) | 0.68 (0.749)
  Q10 (Day 7) | 0.60 (0.883) | 0.60 (0.940) | 0.37 (0.597)
  Q10 (Day 14) | 0.40 (0.754) | 0.55 (0.887) | 0.37 (0.597)
  Q11 (Day 7) | 0.70 (0.801) | 1.30 (0.979) | 1.00 (0.745)
  Q11 (Day 14) | 0.70 (0.865) | 1.05 (0.887) | 0.68 (0.749)
  Q12 (Day 7) | 0.40 (0.754) | 0.70 (0.733) | 0.63 (0.761)
  Q12 (Day 14) | 0.30 (0.733) | 0.60 (0.821) | 0.32 (0.582)
  Q13 (Day 7) | 0.45 (0.605) | 0.70 (0.733) | 0.74 (0.733)
  Q13 (Day 14) | 0.55 (0.605) | 0.60 (0.754) | 0.63 (0.761)
  Q14 (Day 7) | 0.35 (0.489) | 0.65 (0.745) | 0.53 (0.697)
  Q14 (Day 14) | 0.45 (0.605) | 0.55 (0.605) | 0.53 (0.612)
  Q15 (Day 7) | 1.00 (0.324) | 1.20 (0.616) | 1.32 (0.582)
  Q15 (Day 14) | 1.05 (0.394) | 1.05 (0.510) | 1.05 (0.621)
  Q16 (Day 7) | 0.40 (0.754) | 0.74 (0.933) | 0.47 (0.697)
  Q16 (Day 14) | 0.25 (0.716) | 0.50 (0.688) | 0.32 (0.582)
  Q 19 (Day 7) | 1.40 (0.754) | 2.00 (0.795) | 1.68 (0.671)
  Q19 (Day 14) | 1.35 (0.587) | 1.70 (0.865) | 1.26 (0.733)
  Q20 (Day 7) | 1.30 (0.923) | 1.85 (0.933) | 1.63 (0.684)
  Q20 (Day 14) | 1.40 (0.821) | 1.75 (0.967) | 1.21 (0.713)

16. Secondary Outcome: Summary of Other Daily Diary VAS Scale Questions Before and After Strip Application at Bedtime
Description: Participants were asked how easy it was to breathe through their nose before and after strip application at bedtime. The participants scored their responses on VAS scale where 0 = extremely difficult to breathe and 100 = extremely easy to breathe. These responses were recorded daily.
Time Frame: At Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 8, Day 9, Day 10, Day 11, Day 12, and Day 13
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a scale
  Before strip application (Day 1): number analyzed (Participants) | 20 | 19 | 19
  Before strip application (Day 1) | 27.85 (20.582) | 34.58 (15.798) | 34.00 (14.821)
  After strip application (Day 1): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 1) | 61.55 (26.716) | 43.11 (24.071) | 55.00 (24.866)
  Before strip application (Day 2): number analyzed (Participants) | 20 | 19 | 19
  Before strip application (Day 2) | 28.2 (20.18) | 37.2 (23.18) | 42.7 (19.26)
  After strip application (Day 2): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 2) | 60.1 (26.16) | 45.2 (25.04) | 60.7 (22.36)
  Before strip application (Day 3): number analyzed (Participants) | 20 | 19 | 19
  Before strip application (Day 3) | 29.35 (20.296) | 37.95 (19.842) | 45.11 (23.870)
  After strip application (Day 3): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 3) | 58.90 (26.638) | 48.53 (20.665) | 61.42 (24.739)
  Before strip application (Day 4): number analyzed (Participants) | 20 | 19 | 18
  Before strip application (Day 4) | 32.8 (20.87) | 33.3 (14.27) | 36.4 (19.29)
  After Strip application (Day 4): number analyzed (Participants) | 20 | 19 | 18
  After Strip application (Day 4) | 60.8 (28.86) | 45.7 (17.89) | 60.2 (22.14)
  Before strip application (Day 5): number analyzed (Participants) | 20 | 19 | 19
  Before strip application (Day 5) | 33.2 (23.45) | 36.9 (19.78) | 41.4 (21.85)
  After strip application (Day 5): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 5) | 64.9 (28.11) | 47.5 (22.51) | 63.8 (23.95)
  Before strip application (Day 6): number analyzed (Participants) | 20 | 19 | 19
  Before strip application (Day 6) | 28.6 (22.47) | 35.9 (20.29) | 44.9 (18.55)
  After strip application (Day 6): number analyzed (Participants) | 20 | 18 | 19
  After strip application (Day 6) | 60.5 (30.06) | 44.8 (21.28) | 64.3 (20.03)
  Before strip application (Day 8): number analyzed (Participants) | 20 | 19 | 19
  Before strip application (Day 8) | 35.4 (22.08) | 38.6 (21.38) | 45.5 (19.18)
  After strip application (Day 8): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 8) | 61.2 (26.41) | 47.8 (25.07) | 65.0 (22.96)
  Before strip application (Day 9): number analyzed (Participants) | 20 | 19 | 19
  Before strip application (Day 9) | 32.7 (24.11) | 40.0 (21.18) | 45.6 (19.90)
  After strip application (Day 9): number analyzed (Participants) | 20 | 18 | 19
  After strip application (Day 9) | 61.2 (27.90) | 48.6 (24.45) | 63.4 (22.45)
  Before strip application (Day 10): number analyzed (Participants) | 20 | 19 | 19
  Before strip application (Day 10) | 36.9 (25.80) | 42.7 (27.71) | 40.6 (19.74)
  After strip application (Day 10): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 10) | 68.3 (27.76) | 50.2 (30.15) | 60.9 (24.91)
  After strip application (Day 11): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 11) | 66.3 (26.45) | 49.8 (25.18) | 63.2 (25.60)
  Before strip application (Day 11): number analyzed (Participants) | 20 | 19 | 19
  Before strip application (Day 11) | 33.6 (25.33) | 40.2 (22.99) | 42.1 (21.52)
  Before strip application (Day 12): number analyzed (Participants) | 19 | 19 | 19
  Before strip application (Day 12) | 32.7 (25.79) | 42.5 (24.96) | 47.5 (21.51)
  After strip application (Day 12): number analyzed (Participants) | 19 | 19 | 19
  After strip application (Day 12) | 66.8 (27.43) | 52.8 (26.46) | 65.7 (23.44)
  Before strip application (Day 13): number analyzed (Participants) | 20 | 19 | 19
  Before strip application (Day 13) | 33.9 (27.28) | 43.5 (23.07) | 48.1 (24.12)
  After strip application (Day 13): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 13) | 66.7 (26.62) | 53.1 (26.16) | 67.8 (24.38)

17. Secondary Outcome: Summary of Other Daily Diary VAS Scale Questions Before and After Strip Removal in Morning
Description: Participants were asked how easy it was to breathe through their nose before and after strip removal in morning. The participants scored their responses on VAS scale where 0 = extremely difficult to breathe and 100 = extremely easy to breathe. These responses were recorded daily.
Time Frame: At Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 8, Day 9, Day 10, Day 11, Day 12, and Day 13
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a scale
  Before strip removal (Day 1): number analyzed (Participants) | 20 | 19 | 18
  Before strip removal (Day 1) | 54.60 (30.407) | 45.11 (22.588) | 60.44 (20.024)
  After strip removal (Day 1): number analyzed (Participants) | 20 | 19 | 18
  After strip removal (Day 1) | 44.75 (21.560) | 41.47 (20.018) | 51.44 (20.569)
  Before strip removal (Day 2): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 2) | 61.0 (26.25) | 44.1 (22.56) | 60.0 (22.85)
  After strip removal (Day 2): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 2) | 46.8 (21.80) | 42.1 (22.34) | 51.2 (21.76)
  Before strip removal (Day 3): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 3) | 63.60 (27.582) | 48.37 (23.864) | 60.21 (24.114)
  After strip removal (Day 3): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 3) | 44.90 (21.071) | 45.53 (23.236) | 56.79 (21.578)
  Before strip removal (Day 4): number analyzed (Participants) | 20 | 19 | 18
  Before strip removal (Day 4) | 64.9 (26.35) | 50.0 (19.06) | 62.8 (21.56)
  After strip removal (Day 4): number analyzed (Participants) | 20 | 19 | 18
  After strip removal (Day 4) | 49.2 (23.37) | 45.9 (21.27) | 53.6 (20.99)
  Before strip removal (Day 5): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 5) | 65.0 (27.48) | 47.4 (21.94) | 64.0 (20.90)
  After strip removal (Day 5): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 5) | 49.7 (23.50) | 43.4 (23.21) | 58.1 (19.31)
  Before strip removal (Day 6): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 6) | 60.9 (27.34) | 46.2 (23.94) | 63.1 (21.40)
  After strip removal (Day 6): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 6) | 47.0 (24.03) | 42.4 (23.16) | 58.6 (18.40)
  Before strip removal (Day 8): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 8) | 64.7 (25.34) | 43.6 (25.55) | 65.2 (20.39)
  After strip removal (Day 8): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 8) | 46.6 (25.50) | 40.7 (24.07) | 60.4 (19.35)
  Before strip removal (Day 9): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 9) | 61.1 (27.82) | 46.7 (24.68) | 65.1 (23.06)
  After strip removal (Day 9): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 9) | 49.0 (26.34) | 41.7 (24.08) | 59.5 (20.19)
  Before strip removal (Day 10): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 10) | 66.2 (25.85) | 45.6 (26.88) | 65.4 (22.52)
  After strip removal (Day 10): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 10) | 50.6 (24.92) | 42.4 (26.57) | 57.5 (22.10)
  Before strip removal (Day 11): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 11) | 62.3 (26.37) | 47.3 (25.79) | 67.5 (20.50)
  After strip removal (Day 11): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 11) | 46.4 (23.93) | 42.2 (23.98) | 57.0 (19.91)
  Before strip removal (Day 12): number analyzed (Participants) | 19 | 19 | 19
  Before strip removal (Day 12) | 63.8 (25.58) | 49.2 (24.95) | 67.6 (21.03)
  After strip removal (Day 12): number analyzed (Participants) | 19 | 19 | 19
  After strip removal (Day 12) | 48.7 (27.39) | 46.3 (23.45) | 59.4 (21.30)
  Before strip removal (Day 13): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 13) | 64.3 (25.58) | 46.4 (26.18) | 68.4 (22.84)
  After strip removal (Day 13): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 13) | 46.6 (27.39) | 43.3 (26.37) | 60.0 (21.02)

18. Secondary Outcome: Summary of Other Daily Diary VAS Scale Questions Before and After Strip Application at Bedtime
Description: Participants were asked how open their nose feels before and after strip application at bedtime. The participants scored their responses VAS scale where 0 = nose was extremely blocked and 100 = nose was extremely clear. These responses were recorded daily.
Time Frame: At Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 8, Day 9, Day 10, Day 11, Day 12, and Day 13
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a Scale
  Before strip application (Day 1): number analyzed (Participants) | 20 | 19 | 18
  Before strip application (Day 1) | 27.90 (20.463) | 37.74 (17.143) | 35.89 (14.644)
  After strip application (Day 1): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 1) | 61.45 (25.853) | 45.84 (23.061) | 57.68 (22.583)
  Before strip application (Day 2): number analyzed (Participants) | 20 | 19 | 19
  Before strip application (Day 2) | 27.5 (19.64) | 38.3 (22.17) | 42.2 (19.49)
  After strip application (Day 2): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 2) | 59.8 (26.90) | 47.0 (24.10) | 63.2 (63.2)
  Before strip application (Day 3): number analyzed (Participants) | 20 | 19 | 19
  Before strip application (Day 3) | 30.05 (20.405) | 38.32 (19.285) | 46.42 (24.132)
  After strip application (Day 3): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 3) | 59.25 (27.466) | 49.74 (22.098) | 62.16 (24.847)
  Before strip application (Day 4): number analyzed (Participants) | 20 | 19 | 18
  Before strip application (Day 4) | 32.6 (20.51) | 33.6 (14.78) | 36.6 (18.74)
  After strip application (Day 4): number analyzed (Participants) | 20 | 19 | 18
  After strip application (Day 4) | 60.5 (28.31) | 46.7 (17.34) | 61.1 (23.41)
  Before strip application (Day 5): number analyzed (Participants) | 20 | 19 | 19
  Before strip application (Day 5) | 33.4 (23.85) | 36.1 (19.57) | 42.1 (21.60)
  After strip appliation (Day 5): number analyzed (Participants) | 19 | 19 | 19
  After strip appliation (Day 5) | 65.6 (28.44) | 49.3 (22.62) | 66.7 (23.97)
  Before strip application (Day 6): number analyzed (Participants) | 19 | 19 | 19
  Before strip application (Day 6) | 26.7 (20.58) | 35.3 (18.59) | 44.8 (20.14)
  After strip application (Day 6): number analyzed (Participants) | 20 | 18 | 19
  After strip application (Day 6) | 60.5 (28.86) | 43.9 (19.34) | 66.5 (20.92)
  Before strip application (Day 8): number analyzed (Participants) | 19 | 19 | 18
  Before strip application (Day 8) | 33.9 (21.15) | 37.9 (22.54) | 46.9 (20.76)
  After strip application (Day 8): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 8) | 63.4 (26.94) | 46.5 (24.74) | 67.5 (67.5)
  Before strip application (Day 9): number analyzed (Participants) | 19 | 18 | 19
  Before strip application (Day 9) | 32.7 (24.42) | 37.6 (20.70) | 45.8 (21.77)
  After strip application (Day 9): number analyzed (Participants) | 20 | 18 | 19
  After strip application (Day 9) | 65.6 (26.71) | 49.5 (25.34) | 65.5 (23.09)
  Before strip application (Day 10): number analyzed (Participants) | 20 | 19 | 19
  Before strip application (Day 10) | 36.2 (42.1) | 42.1 (26.94) | 41.8 (22.31)
  After strip application (Day 10): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 10) | 68.7 (26.85) | 52.1 (30.45) | 63.0 (25.34)
  Before strip application (Day 11): number analyzed (Participants) | 20 | 19 | 19
  Before strip application (Day 11) | 35.4 (24.79) | 41.3 (23.74) | 41.3 (22.54)
  After strip application (Day 11): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 11) | 67.3 (26.69) | 50.5 (27.02) | 64.8 (25.15)
  Before strip application (Day 12): number analyzed (Participants) | 18 | 18 | 19
  Before strip application (Day 12) | 34.7 (26.71) | 44.2 (24.78) | 47.5 (23.30)
  After strip application (Day 12): number analyzed (Participants) | 19 | 19 | 19
  After strip application (Day 12) | 68.4 (26.67) | 53.4 (26.40) | 67.5 (23.95)
  Before strip application (Day 13): number analyzed (Participants) | 20 | 19 | 19
  Before strip application (Day 13) | 34.9 (26.36) | 42.7 (23.58) | 50.3 (24.75)
  After strip application (Day 13): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 13) | 67.1 (25.90) | 53.6 (25.74) | 68.1 (25.28)

19. Secondary Outcome: Summary of Other Daily Diary VAS Scale Questions Before and After Strip Removal in Morning.
Description: Participants were asked how open their nose feels before and after strip removal in morning. The participants scored their responses VAS scale where 0 = nose was extremely blocked and 100 = nose was extremely clear. These responses were recorded daily.
Time Frame: At Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 8, Day 9, Day 10, Day 11, Day 12, and Day 13
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Prototype Nasal Strip: Participants applied the Prototype nasal dilator strips according to written instructions to be provided. A member of the site staff reviewed the instructions for administration with each participant. Strips were applied every night during the treatment phase of the study. All treatments in this study were self-administered by the participant.
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a Scale
  Before strip removal (Day 1): number analyzed (Participants) | 20 | 19 | 18
  Before strip removal (Day 1) | 53.95 (29.883) | 45.37 (25.049) | 60.22 (21.198)
  After strip removal (Day 1): number analyzed (Participants) | 20 | 19 | 18
  After strip removal (Day 1) | 44.70 (22.181) | 42.53 (20.291) | 51.56 (22.727)
  Before strip removal (Day 2): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 2) | 60.8 (26.46) | 43.7 (20.85) | 60.6 (23.48)
  After strip removal (Day 2): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 2) | 45.7 (23.56) | 43.4 (22.56) | 53.1 (22.81)
  Before strip removal (Day 3): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 3) | 61.35 (27.871) | 46.89 (23.812) | 60.53 (24.688)
  After strip removal (Day 3): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 3) | 44.30 (21.440) | 45.47 (22.473) | 58.11 (22.652)
  Before strip removal (Day 4): number analyzed (Participants) | 20 | 19 | 18
  Before strip removal (Day 4) | 63.7 (25.51) | 48.2 (19.23) | 64.7 (22.55)
  After strip removal (Day 4): number analyzed (Participants) | 20 | 19 | 17
  After strip removal (Day 4) | 48.3 (22.10) | 45.5 (21.18) | 55.1 (21.13)
  Before strip removal (Day 5): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 5) | 65.2 (27.66) | 45.2 (23.74) | 64.4 (20.52)
  After strip removal (Day 5): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 5) | 49.3 (25.08) | 43.4 (23.30) | 59.6 (20.14)
  Before strip removal (Day 6): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 6) | 60.4 (27.25) | 45.9 (24.34) | 64.9 (22.29)
  After strip removal (Day 6): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 6) | 45.0 (22.74) | 45.6 (22.77) | 58.8 (19.74)
  Before strip removal (Day 8): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 8) | 65.3 (25.65) | 41.6 (25.54) | 66.7 (21.14)
  After strip removal (Day 8): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 8) | 46.9 (26.82) | 42.5 (24.62) | 59.7 (19.85)
  Before strip removal (Day 9): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 9) | 62.8 (25.86) | 43.3 (24.41) | 65.5 (21.99)
  After strip removal (Day 9): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 9) | 48.3 (27.55) | 40.1 (24.98) | 60.2 (20.34)
  Before strip removal (Day 10): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 10) | 66.1 (25.67) | 43.1 (26.52) | 67.1 (23.01)
  After strip removal (Day 10): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 10) | 50.6 (25.43) | 42.7 (26.55) | 57.6 (22.72)
  Before strip removal (Day 11): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 11) | 61.6 (26.54) | 44.3 (25.67) | 67.2 (21.63)
  After strip removal (Day 11): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 11) | 47.1 (23.92) | 42.2 (24.54) | 24.54 (20.87)
  Before strip removal (Day 12): number analyzed (Participants) | 19 | 19 | 19
  Before strip removal (Day 12) | 63.1 (26.12) | 46.5 (23.72) | 69.2 (20.81)
  After strip removal (Day 12): number analyzed (Participants) | 19 | 19 | 19
  After strip removal (Day 12) | 49.7 (27.52) | 47.4 (21.72) | 61.8 (22.26)
  Before strip removal (Day 13): number analyzed (Participants) | 20 | 18 | 19
  Before strip removal (Day 13) | 64.9 (25.41) | 40.9 (24.83) | 68.6 (22.41)
  After strip removal (Day 13): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 13) | 46.4 (28.24) | 42.3 (24.85) | 61.0 (22.33)

20. Secondary Outcome: Summary of Daily Diary Questions Before and After Strip Application at Bedtime
Description: Participants were asked how stuffed their nose felt before and after strip application at bed time. The participants scored their responses on the scale of 0 to 3 where 0=No symptoms, 1=mild symptoms and 3=severe symptoms. These responses were recorded daily.
Time Frame: At Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 8, Day 9, Day 10, Day 11, Day 12, and Day 13
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a scale
  Before strip application (Day 1) | 1.95 (0.394) | 2.00 (0.562) | 1.79 (0.535)
  After strip application (Day 1) | 1.10 (0.788) | 1.80 (0.696) | 1.26 (0.562)
  Before strip application (Day 2) | 1.80 (0.696) | 1.85 (0.587) | 1.53 (0.612)
  After strip application (Day 2) | 1.05 (0.686) | 1.70 (0.733) | 1.11 (0.658)
  Before strip application (Day 3) | 1.90 (0.641) | 1.90 (0.553) | 1.58 (0.692)
  After strip application (Day 3): number analyzed (Participants) | 19 | 20 | 19
  After strip application (Day 3) | 1.16 (0.898) | 1.60 (0.754) | 1.16 (0.688)
  Before strip application (Day 4) | 1.55 (0.686) | 1.70 (0.733) | 1.74 (0.562)
  After strip application (Day 4) | 0.95 (0.887) | 1.55 (0.759) | 1.16 (0.602)
  Before strip application (Day 5) | 1.75 (0.550) | 1.65 (0.671) | 1.53 (0.772)
  After strip application (Day 5) | 1.00 (0.795) | 1.50 (0.761) | 1.21 (0.855)
  Before strip application (Day 6) | 1.90 (0.641) | 1.75 (0.716) | 1.53 (0.697)
  After strip application (Day 6) | 1.00 (0.795) | 1.65 (0.813) | 1.16 (0.501)
  Before strip application (Day 8) | 1.70 (0.571) | 1.70 (0.571) | 1.47 (0.513)
  After strip application (Day 8): number analyzed (Participants) | 20 | 19 | 18
  After strip application (Day 8) | 1.15 (0.813) | 1.47 (0.772) | 0.83 (0.786)
  Before strip application (Day 9): number analyzed (Participants) | 20 | 19 | 18
  Before strip application (Day 9) | 1.70 (0.571) | 1.58 (0.838) | 1.39 (0.608)
  After strip application (Day 9): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 9) | 1.05 (0.826) | 1.37 (0.955) | 1.05 (0.705)
  Before strip application (Day 10) | 1.60 (0.598) | 1.65 (0.933) | 1.37 (0.831)
  After strip application (Day 10) | 0.95 (0.945) | 1.50 (1.051) | 1.21 (0.918)
  Before strip application (Day 11): number analyzed (Participants) | 19 | 20 | 18
  Before strip application (Day 11) | 1.68 (0.671) | 1.60 (0.821) | 1.56 (0.616)
  After strip application (Day 11): number analyzed (Participants) | 20 | 20 | 18
  After strip application (Day 11) | 1.15 (0.875) | 1.45 (0.945) | 1.11 (0.676)
  Before strip application (Day 12): number analyzed (Participants) | 19 | 20 | 19
  Before strip application (Day 12) | 1.74 (0.653) | 1.40 (0.754) | 1.37 (0.684)
  After strip application (Day 12): number analyzed (Participants) | 19 | 19 | 19
  After strip application (Day 12) | 1.05 (0.911) | 1.26 (0.872) | 0.95 (0.621)
  Before strip application (Day 13): number analyzed (Participants) | 20 | 20 | 18
  Before strip application (Day 13) | 1.75 (0.639) | 1.50 (0.688) | 1.39 (0.850)
  After strip applications (Day 13) | 0.90 (0.912) | 1.35 (0.813) | 1.05 (0.848)

21. Secondary Outcome: Summary of Daily Dairy Questions Before and After Strip Removal in Morning
Description: Participants were asked how stuffed their nose felt before and after strip removal in morning. The participants scored their responses on the scale of 0 to 3 where 0=No symptoms, 1=mild symptoms and 3=severe symptoms. These responses were recorded daily.
Time Frame: At Day 1, Day 2, day 3, Day 4, Day 5, Day 6, Day 8, Day 9, Day 10, Day 11, Day 12, and Day 13
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a scale
  Before strip removal (Day 1): number analyzed (Participants) | 20 | 20 | 18
  Before strip removal (Day 1) | 1.15 (0.745) | 1.55 (0.759) | 1.22 (0.647)
  After strip removal (Day 1): number analyzed (Participants) | 20 | 20 | 18
  After strip removal (Day 1) | 1.35 (0.671) | 1.65 (0.745) | 1.33 (0.594)
  Before strip removal (Day 2): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 2) | 1.05 (0.686) | 1.53 (0.905) | 1.21 (0.855)
  After strip removal (Day 2) | 1.40 (0.681) | 1.70 (0.801) | 1.32 (0.671)
  Before strip removal (Day 3): number analyzed (Participants) | 19 | 20 | 19
  Before strip removal (Day 3) | 0.84 (0.688) | 1.45 (0.887) | 1.11 (0.737)
  After strip removal (Day 3): number analyzed (Participants) | 20 | 20 | 18
  After strip removal (Day 3) | 1.35 (0.671) | 1.55 (0.826) | 1.11 (0.583)
  Before strip removal (Day 4): number analyzed (Participants) | 20 | 19 | 19
  Before strip removal (Day 4) | 0.95 (0.826) | 1.42 (0.838) | 1.00 (0.816)
  After strip removal (Day 4) | 1.25 (0.639) | 1.55 (0.759) | 1.11 (0.658)
  Before strip removal (Day 5) | 0.95 (0.759) | 1.40 (0.821) | 1.00 (0.882)
  After strip removal (Day 5) | 1.25 (0.786) | 1.55 (0.826) | 0.95 (0.621)
  Before strip removal (Day 6) | 1.05 (0.826) | 1.55 (0.999) | 1.00 (0.816)
  After strip removal (Day 6) | 1.40 (0.754) | 1.65 (0.933) | 1.05 (0.621)
  Before strip removal (Day 8) | 1.05 (0.759) | 1.55 (0.945) | 0.84 (0.688)
  After strip removal (Day 8): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 8) | 1.45 (0.826) | 1.68 (0.885) | 1.00 (0.745)
  Before strip removal (Day 9) | 0.95 (0.826) | 1.45 (1.050) | 0.79 (0.631)
  After strip removal (Day 9): number analyzed (Participants) | 20 | 19 | 19
  After strip removal (Day 9) | 1.45 (0.826) | 1.58 (1.017) | 0.95 (0.621)
  Before strip removal (Day 10): number analyzed (Participants) | 20 | 20 | 18
  Before strip removal (Day 10) | 0.90 (0.852) | 1.60 (0.995) | 1.00 (0.767)
  After strip removal (Day 10) | 1.20 (0.768) | 1.60 (0.940) | 1.21 (0.713)
  Before strip removal (Day 11) | 1.20 (0.834) | 1.55 (0.945) | 1.00 (0.577)
  After strip removal (Day 11) | 1.50 (0.761) | 1.70 (0.923) | 1.21 (0.631)
  Before strip removal (Day 12): number analyzed (Participants) | 19 | 20 | 19
  Before strip removal (Day 12) | 1.00 (0.882) | 1.30 (1.031) | 0.74 (0.733)
  After strip removal (Day 12): number analyzed (Participants) | 19 | 20 | 19
  After strip removal (Day 12) | 1.37 (0.831) | 1.40 (0.995) | 0.95 (0.621)
  Before strip removal (Day 13) | 0.95 (0.826) | 1.50 (1.000) | 1.00 (0.745)
  After strip removal (Day 13) | 1.40 (0.883) | 1.65 (0.933) | 1.05 (0.848)

22. Secondary Outcome: Summary of Daily Diary Questions at Bed Time (After Strip Application) and in Morning (After Strip Removal).
Description: Participants were asked how breathing felt after nasal strip was applied at bed time and removed in morning. The participants scored their responses on the scale of -5 to 5 where -5 = much worse, 0 = same and 5= much better. These responses were recorded daily.
Time Frame: At Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 8, Day 9, Day 10, Day 11, Day 12, and Day13
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a scale
  After strip application (Day 1) | 2.45 (1.395) | 1.20 (1.473) | 1.42 (2.116)
  After strip removal (Day 1): number analyzed (Participants) | 20 | 20 | 18
  After strip removal (Day 1) | -0.30 (2.055) | 0.25 (1.650) | 0.50 (2.407)
  After strip application (Day 2) | 1.95 (1.932) | 0.90 (1.410) | 1.53 (1.744)
  After strip removal (Day 2) | -0.10 (2.075) | 0.30 (1.525) | 0.26 (2.182)
  After strip application (Day 3) | 2.40 (1.667) | 1.20 (1.361) | 1.74 (1.727)
  After strip removal (Day 3) | -0.35 (2.183) | 0.85 (1.631) | 0.68 (1.734)
  After strip application (Day 4) | 2.70 (1.525) | 1.10 (1.334) | 1.47 (1.896)
  After strip removal (Day 4) | -0.50 (2.115) | 0.45 (1.731) | 0.47 (2.118)
  After strip application (Day 5) | 2.80 (1.765) | 1.05 (1.605) | 1.63 (1.707)
  After strip removal (Day 5) | -0.20 (2.397) | 0.55 (1.731) | 0.84 (2.167)
  After strip application (Day 6) | 2.85 (1.565) | 0.95 (1.504) | 1.89 (1.629)
  After strip removal (Day 6) | -0.45 (2.282) | 0.50 (1.792) | 0.74 (2.077)
  After strip application (Day 8) | 2.65 (1.755) | 0.85 (1.309) | 1.84 (1.864)
  After strip removal (Day 8) | -0.45 (2.164) | 0.25 (1.164) | 0.79 (2.043)
  After strip application (Day 9): number analyzed (Participants) | 20 | 19 | 19
  After strip application (Day 9) | 2.80 (1.576) | 0.84 (1.344) | 1.84 (1.675)
  After strip removal (Day 9) | -0.40 (2.415) | 0.20 (1.196) | 1.00 (1.856)
  After strip application (Day 10) | 2.85 (1.599) | 0.95 (1.234) | 1.95 (1.580)
  After strip removal (Day 10): number analyzed (Participants) | 19 | 20 | 19
  After strip removal (Day 10) | -0.47 (2.412) | 0.25 (1.251) | 1.00 (2.082)
  After strip application (Day 11) | 2.60 (1.759) | 0.75 (1.293) | 1.84 (1.675)
  After strip removal (Day 11) | -0.65 (2.277) | 0.10 (1.410) | 0.68 (2.056)
  After strip application (Day 12): number analyzed (Participants) | 19 | 20 | 19
  After strip application (Day 12) | 2.79 (1.782) | 0.95 (1.317) | 2.00 (1.491)
  After strip removal (Day 12): number analyzed (Participants) | 19 | 20 | 19
  After strip removal (Day 12) | -0.74 (2.306) | 0.30 (1.218) | 0.89 (2.052)
  After strip application (Day 13) | 2.65 (1.631) | 0.95 (1.317) | 2.05 (1.649)
  After strip removal (Day 13) | -0.40 (2.703) | 0.35 (1.424) | 0.79 (1.988)

23. Secondary Outcome: Change From Baseline in Mean Average Score of NRQLQ for Each Domain (Sleep, Sleep Time, Symptoms on Waking in the Morning, and Practical Problems) on the) at Day 7 and Day 14 in Participants With the Risk of Sleep Apnea.
Description: as for outcome 4
Time Frame: At Day 7 and at Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Score on a scale
  Sleep Problems (Day 7): number analyzed (Participants) | 13 | 12 | 11
  Sleep Problems (Day 7) | 7.62 (6.117) | 11.58 (7.452) | 6.09 (4.826)
  Sleep Problems (Day 14): number analyzed (Participants) | 13 | 12 | 11
  Sleep Problems (Day 14) | 6.92 (5.951) | 9.75 (6.771) | 4.91 (4.134)
  Sleep time problems (Day 7): number analyzed (Participants) | 13 | 12 | 11
  Sleep time problems (Day 7) | 7.62 (6.838) | 10.08 (7.489) | 6.00 (7.225)
  Sleep time problems (Day 14): number analyzed (Participants) | 13 | 12 | 11
  Sleep time problems (Day 14) | 6.77 (7.683) | 8.50 (8.713) | 6.18 (7.054)
  Symptoms on waking in morning (Day 7): number analyzed (Participants) | 13 | 12 | 11
  Symptoms on waking in morning (Day 7) | 8.69 (6.701) | 12.00 (5.673) | 5.45 (4.228)
  Symptoms on waking in morning (Day 14): number analyzed (Participants) | 13 | 12 | 11
  Symptoms on waking in morning (Day 14) | 8.31 (5.936) | 10.42 (6.543) | 5.00 (4.472)
  Practical problems (Day 7): number analyzed (Participants) | 13 | 12 | 11
  Practical problems (Day 7) | 3.00 (5.033) | 4.67 (3.601) | 2.55 (3.503)
  Practical Problems (Day 14): number analyzed (Participants) | 13 | 12 | 11
  Practical Problems (Day 14) | 2.54 (4.858) | 3.08 (3.059) | 2.64 (2.942)

24. Secondary Outcome: Number of Participants Showing Improvement for Sleep Problems and Symptoms on Waking in the Morning Domain of the NRQLQ
Description: Participants scored all two domains of NRQLQ using same 7 points scale: 0=Not troubled, 1=Hardly troubled, 3=moderately troubled, 4=quite a bit troubled, 5=very troubled, 6=extremely troubled. Domains were Sleep problems (difficulty getting sleep, unable to get a good night sleep or wake up during the night, restless [tossing and turning] and having to get up because stuffy nose or to blow nose using the score), and Symptoms on waking in the morning (Feel tired and unrefreshed, nasal congestion or stuffy nose, congestion in sinuses, takes time to clear nighttime drainage after waking up); Lower scores indicate improvement in the rhinitis symptoms.
Time Frame: At Day 7 and Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Participants
  All sleep problems (Day 7) | 14 | 5 | 11
  All sleep problems (Day 14) | 12 | 10 | 13
  Any sleep problems (Day 7) | 18 | 18 | 19
  Any sleep problems (Day 14) | 20 | 19 | 17
  All symptoms on waking (Day 7) | 14 | 11 | 14
  All symptoms on waking (Day 14) | 14 | 11 | 16
  Any symptoms on waking (Day 7) | 19 | 17 | 19
  Any symptoms on waking (Day 14) | 19 | 18 | 19

25. Secondary Outcome: Number of Participants Showing Improvement for Daily Diary Questions (Q2 and Q4)
Description: Participants were asked Q2 (How stuffed does your nose feel at this time?) and Q4 (How Breathing felt after the nasal strip was applied) of daily diary questions. Q2 was scored on 4 point scale where 0=no symptoms, 1=mild symptoms, 2=moderate symptoms, 3=severe symptoms and Q4 on 11 point scale where -5=much worse, 0=same, 5=much better.
Time Frame: on first night (Night 1) of each daily diary question
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Participants
  Q2 | 13 | 3 | 10
  Q4 | 18 | 11 | 12

26. Secondary Outcome: Number of Participants Showing Improvement for VAS Scale Daily Diary Questions
Description: Participants were asked following daily diary VAS scale questions a) How easy it was to breathe through your nose and b) How open their nose feels at this time. Both of these questions were scored using 100 mm VAS scale where, 0=extremely difficult, 100=extremely easy.
Time Frame: on first night (Night 1) of each daily diary question
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Strip
Number analyzed (Participants) | 20 | 20 | 19
Participants
  Easy to breathe | 20 | 11 | 15
  Openness | 19 | 13 | 13

ADVERSE EVENTS:
Groups:
- Prototype Nasal Dilator: Participants applied the Prototype nasal strips according to written instructions. A member of the site staff reviewed the instructions for administration with each participant. Strips were applied every night during the treatment phase of the study. All treatments in this study were self-administered by the participant.
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Prototype Nasal Dilator
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 1/21 | 0/19
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Marketed Nasal Strip (N=20) | Placebo Nasal Strip (N=21) | Prototype Nasal Dilator (N=19)
Nasal scab secondary to strip removal (General disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.